CLINICAL TRIAL: NCT00677144
Title: A Randomized Phase II Study of Oxaliplatin and S-1 (OS) Versus Oxaliplatin and Capecitabine (XELOX) in Patients With Advanced or Recurrent Colorectal Cancer
Brief Title: Oxaliplatin and S-1 (OS) Versus Oxaliplatin and Capecitabine (XELOX) for Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMC-HO-GI-0712
Record Dates: First submitted 2008-05-07; First posted 2008-05-13 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Colorectal Neoplasm
Keywords: Colorectal Neoplasm; S-1; Capecitabine; Oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; titanium silicide; XELOX; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OS (oxalipaltin+S-1) (Experimental): OS (oxaliplatin + S-1): Oxaliplatin 130mg/m2 IV on D1 every 21 days and S-1 80mg/m2/day PO [BSA <1.25 40mg bid (total 80mg/day); BSA ≥1.25 - <1.5 50mg bid (total 100mg/day); BSA ≥1.5 60mg bid (total 120mg/day)], divided by two on D1-14 every 21 days
  Interventions: Drug: OS (oxalipaltin+S-1)
- XELOX (oxalipaltin+capecitabine) (Active Comparator): XELOX (oxalipaltin+capecitabine): Oxaliplatin 130mg/m2 IV on D1 every 21 days and Capecitabine 2000mg/m2/day PO, divided by two on D1-14 every 21 days
  Interventions: Drug: XELOX (oxalipaltin+capecitabine)

INTERVENTIONS:
Drug: OS (oxalipaltin+S-1) — Oxaliplatin 130mg/m2 IV on D1 every 21 days and S-1 80mg/m2/day PO [BSA <1.25 40mg bid (total 80mg/day); BSA ≥1.25 - <1.5 50mg bid (total 100mg/day); BSA ≥1.5 60mg bid (total 120mg/day)], divided by two on D1-14 every 21 days
  Other Names: Eloxatin; TS-1
  Arms: OS (oxalipaltin+S-1)
Drug: XELOX (oxalipaltin+capecitabine) — Oxaliplatin 130mg/m2 IV on D1 every 21 days and Capecitabine 2000mg/m2/day PO, divided by two on D1-14 every 21 days
  Other Names: Eloxatin; Xeloda
  Arms: XELOX (oxalipaltin+capecitabine)

SUMMARY:
The aim of this study is to compare the activity and safety of Oxaliplatin and S-1 (OS) and Oxaliplatin and Capecitabine (XELOX) in patients with advance or recurrent colorectal cancer.

DETAILED DESCRIPTION:
Oxaliplatin and oral fluoropyrimidines (capecitabine or S-1) are active agents for colorectal cancer. Recent a phase II trial of combination chemotherapy of oxaliplatin with S-1 (OS) and several phase II trial of combination chemotherapy of oxaliplatin with capecitabine (XELOX) demonstrated good activity and mild toxicity in advanced colorectal cancer. Oxaliplatin and S-1 or capecitabine have distinct mechanisms of action and no overlap of key toxicities. Furthermore, oxaliplatin and fluorouracil were shown to be highly synergistic, not only in preclinical models but also in subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma, initially diagnosed or recurred
* Unresectable, locally advanced or metastatic
* At least one uni-dimensional measurable lesion by RECIST criteria
* Age 18 to 75 years old
* Estimated life expectancy ≥3 months
* ECOG performance status ≤2
* Adequate bone marrow function (WBCs ≥ 4,000/µL or absolute neutrophil count ≥ 1,500/µL, platelets ≥ 100,000/µL)
* Adequate kidney function (creatinine < 1.5 mg/dL)
* Adequate liver function (bilirubin < 2.0 mg/dL, transaminase levels <2.5 times the upper normal limit)
* Written informed consent

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* Previous history of chemotherapy (exception : neoadjuvant or adjuvant chemotherapy without oxaliplatin)
* Presence of CNS metastasis, psychosis, or seizure
* Obvious bowel obstruction
* Evidence of serious gastrointestinal bleeding
* Past or concurrent history of neoplasm other than colorectal adenocarcinoma, except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix uteri
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
overall response rate | 4 years

SECONDARY OUTCOMES:
Safety, time to progression, and overall survival | 4.6 years

CONTACTS AND LOCATIONS:
Overall Officials: Dae Young Zang, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Medical Center, Anyang, South Korea